CLINICAL TRIAL: NCT01267344
Title: A Randomized Phase II Study of Gemcitabine Plus Oxaliplatin (GEMOX) With or Without Cetuximab in Locally Advanced and Metastatic Biliary Tract Cancer (BTC)
Brief Title: A Randomized Study of GEMOX With or Without Cetuximab in Locally Advanced and Metastatic BTC
Acronym: BTC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Mackay Memorial Hospital (Other); Tri-Service General Hospital (Other); Chang Gung Memorial Hospital (Other); Taichung Veterans General Hospital (Other); China Medical University Hospital (Other); National Cheng-Kung University Hospital (Other); Kaohsiung Medical University (Other); Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T1210
Record Dates: First submitted 2010-12-14; First posted 2010-12-28 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2013-10

CONDITIONS: Cholangiocarcinoma; Adenocarcinoma of Gallbladder
Keywords: biliary tract cancer; BTC; cetuximaba
MeSH Terms: conditions — Cholangiocarcinoma; Biliary Tract Neoplasms | interventions — gemcitabine-oxaliplatin regimen; Oxaliplatin; Cetuximab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GEMOX (Active Comparator): Intravenous infusion of gemcitabine 800 mg/m2 at a fixed rate of 10 mg/m2/min followed by oxaliplatin 85 mg/m2 2-hour infusion, every 2 weeks.
  Interventions: Drug: gemcitabine, oxaliplatin
- E-GEMOX (Experimental): Arm A will receive E-GEMOX with additional intravenous infusion of cetuximab (120 minutes for the 1st, 90 minutes for the 2nd and 60 minutes for all subsequent infusions) before GEMOX will be administered as above.
  Interventions: Drug: cetuximab, gemcitabine, oxaliplatin

INTERVENTIONS:
Drug: gemcitabine, oxaliplatin — GEMOX (intravenous infusion of gemcitabine 800 mg/m2 at a fixed rate of 10 mg/m2/min followed by oxaliplatin 85 mg/m2 2-hour infusion, every 2 weeks
  Other Names: Gemmis, Eloxatin
  Arms: GEMOX
Drug: cetuximab, gemcitabine, oxaliplatin — E-GEMOX: intravenous infusion of cetuximab (120 minutes for the 1st, 90 minutes for the 2nd and 60 minutes for all subsequent infusions) before GEMOX will be administered as above. All of the study medication will be administrated on day 1 every 2 weeks, which is regarded as one cycle.
  Other Names: Erbitux@, Eloxatin
  Arms: E-GEMOX

SUMMARY:
The primary objective is to investigate the objective response rate in patients receiving GEMOX (gemcitabine plus oxaliplatin) plus cetuximab as first line treatment in advanced or metastatic unresectable BTC biliary tract cancer compared to patients receiving the same chemotherapy without cetuximab. The secondary objectives include the exploration of the effect of the multimodality strategy on progression-free and overall survival, biomarker prediction, and toxicity.

DETAILED DESCRIPTION:
It is considered realistic, that within 18 months 120 patients can be included in the participating centers. Based on the previous publications an objective response rate (ORR) of 20% is expected in the GEMOX arm (Arm B). When the sample size of evaluable patients is between 110 and 120 evaluable patients (ie. 55 to 60 patients per treatment arm), then a two-sided 95% confidence interval (CI) for the difference between an arm B response rate PB, of 20% and an arm A response rate PA of 30%, 35% or 40% based on the large sample normal approximation will have a width between 15.4% and 16.7%. We assume an objective response rate of 30% for Arm A, then a two-sided 95% confidence interval (CI) for the difference between an arm B response rate PB, of 20% and an arm A response rate PA of 30% will have a width ±15.4% when the sample size of evaluable patients is 120 (i.e., 60 patients per treatment arm).

ELIGIBILITY:
Inclusion criteria:

* Cyto-/histological confirmed unresectable, locally advanced, or metastatic biliary tract cancer, including intrahepatic or extrahepatic cholangiocarcinoma or adenocarcinoma of gallbladder, but NOT other peri-ampulla Vateri or mixed tumor.
* At least one, not previously irradiated, measurable lesion according to RECIST (version 1.1).
* Eastern Cooperative Oncology Group (ECOG) performance score of 0-1.
* Aged no less than 20 years, at the time of acquisition of informed consent.
* Life expectancy >= 3 months.
* Adequate organ and bone marrow function as defined below: WBC >= 3.00 × 103/L and absolute neutrophil count >= 1.50 × 103/L, Platelet count >= 100 × 103/L, Hemoglobin level >= 10 g/dL, Serum creatinine <= 1.5 x Upper Normal Limit (UNL) and calculated GFR >= 40mL/min, Serum bilirubin <= 1.5 x UNL , ALT <= 2.5x UNL.
* Ability to understand and willingness to sign written Informed Consent Form.

Exclusion criteria:

* Other anti-tumor agent such as systemic chemotherapy, immunotherapy or EGFR/VEGF-pathway-targeting therapy before the commencement of study treatment.
* Radiotherapy (except palliative irradiation of bone lesions) within 4 weeks before the commencement of study treatment.
* Other cancer or prior treatment for other carcinomas within the last five years, except cured non-melanoma skin cancer and treated in-situ cervical cancer.
* Known CNS metastasis.
* Major surgery within 4 weeks prior to start of study treatment (diagnostic biopsy, laparotomy, line placement is not considered as major surgery).
* Pre-existing peripheral neuropathy >= grade 2.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, myocardial infarction in the past 12 months, active gastrointestinal bleeding, central nervous system disorders or psychiatric illness/social situation that would limit compliance with study requirements or judged to be ineligible for the study by the investigator.
* Having received any investigational agents or participated in any investigational drug study within 4 weeks prior to study enrollment.
* Pregnant or breast-feeding female (a pregnancy test must be performed on all female patients who are of child-bearing potential before entering the study, and the result must be negative).
* Poor compliance.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
objective response rate | baseline and every 8 weeks
  Evaluation of tumor response according to RECIST 1.1 version Evaluation will be done at baseline and every 8 weeks. Evaluation will be performed with CT or MRI.

SECONDARY OUTCOMES:
The toxicity profiles of the combination treatments | Baseline and every 2 weeks,
  Treatment toxicity will be graded by NCI Common Toxicity Criteria Version 4.0 (CTC, v4.0) for safety evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Li Tz Chen, PHD, Study Chair — National Institute of Cancer Research; Tsang Wu Liu, MD, Study Director — National Institute of Cancer Research, TCOG
Locations (1):
- National Institute of Cancer Research, Taiwan Cooperative Oncology Group, Zhunan, Miaoli County, Taiwan

REFERENCES:
- [Derived] Chen JS, Hsu C, Chiang NJ, Tsai CS, Tsou HH, Huang SF, Bai LY, Chang IC, Shiah HS, Ho CL, Yen CJ, Lee KD, Chiu CF, Rau KM, Yu MS, Yang Y, Hsieh RK, Chang JY, Shan YS, Chao Y, Chen LT; Taiwan Cooperative Oncology Group. A KRAS mutation status-stratified randomized phase II trial of gemcitabine and oxaliplatin alone or in combination with cetuximab in advanced biliary tract cancer. Ann Oncol. 2015 May;26(5):943-949. doi: 10.1093/annonc/mdv035. Epub 2015 Jan 28. PMID 25632066